CLINICAL TRIAL: NCT05794815
Title: Modulation of Gut Microbiota by Probiotic in Children With Respiratory Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: National University of Malaysia (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKMPPI/111/6/JEP-2023-074
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Infection (for Example, Pneumonia, Bronchitis)
Keywords: probiotic; respiratory tract infections; Bifidobacterium; children
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Bronchitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Bifidobacterium infantis YLGB-1496 at 1x10 log CFU/day for 12 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g of maltodextrin, administered daily for 12-weeks)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Bifidobacterium infantis YLGB-1496 at 1x10 log CFU/day for 12 weeks
  Arms: Probiotic
Dietary Supplement: Placebo — Intervention consists of daily administration of 2g of maltodextrin, administered daily for 12-weeks)
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Bifidobacterium infantis YLGB-1496 in modulating gut microbiota of children with respiratory symptoms, among pre-school children in Malaysia aged >12 months old, <7 years old.

DETAILED DESCRIPTION:
Probiotic can be defined as "live microorganisms that grant health effects to the host if consumed in sufficient amounts". Probiotic bacteria, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases.

Respiratory illnesses are the most common acute diseases in children where no virtually effective treatments or prophylaxes are available for these infections. Probiotics on the other hand have gained increasing evidences as an effective therapy in preventing respiratory tract infections. Children attending day care are especially at risk for acquiring respiratory illness, as close physical contact among children in day care favour the transmission of infectious diseases. When studying children receiving either probiotic in milk and control milk, the number of absences from day care because of illness is significantly lesser in probiotic group when compared with control group. In addition, children in the probiotic group had fewer respiratory tract infections with complications (otitis media, sinusitis, bronchitis and pneumonia) and less prescribed antibiotic treatments. The time without respiratory symptoms was also significantly longer in the probiotic group compared with the control group. When the effects of probiotics were studied on nasopharyngeal carriage of bacterial pathogens, the number of human bocavirus was reduced significantly in the nasopharynx of these children, indicating that probiotics may be more effective against respiratory tract infections of viral origin. While the precise mechanisms of using probiotics in management of respiratory infections are largely unknown, speculations include: probiotics compete against pathogens; increase the barrier function in respiratory epithelium; immunostimulatory effects by enhancing cellular immunity with increased activity of natural killer cells and macrophages in airways. Hence, probiotics may offer safe means of reducing the risk of early respiratory related illnesses, common cold and antibiotic use, and the risk of recurrent respiratory infections, thereby represent a simple, safe, effective, available and affordable method for preventing respiratory infections in children.

In worldwide, it is estimated that 5.2 million of children under five of age die every year due to preventable disease such as diarrhea, malaria and pneumonia. Up to date, diarrhea still remains as global health issues, even in developing countries, with 1 million of children deaths reported to be attributed to diarrhea. In Malaysia, reported cases of diarrhea and acute gastroenteritis have been observed to occur throughout the year, with rotavirus-associated diarrhea being the most prevalently identified gastrointestinal disorder. One of the most common gastrointestinal disorders in young children, is diarrhea. Diarrhea is commonly defined as three or more loose or watery stools in the last 24 hours. For clinical studies employing oral administration of probiotics, the probiotics were administered directly to the participants or mixed with a variety of fluids and foods. In studies on probiotic prevention of acute diarrhea in daycare centres worldwide, probiotics tested such as Lactobacillus GG, Bifidobacterium lactis (alone or in combination with Streptococcus thermophiles), and Lactobacillus reuteri, Lactobacillus casei and Lactobacillus acidophilus showed a clear evidence of efficacy to reduce diarrhea-related symptoms in a strain-dependent and dose-dependent manner. Probiotics administration reduces duration of diarrhea, indicating the efficacy of probiotics not only in preventing occurrence of diarrhea, as well as to treat episodes of diarrhea. Probiotics Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium longum and Saccharomyces boulardii also showed decreased time of vomiting in the intervention groups as compared with controls during the probiotics treatment of acute rotavirus diarrhoea. The rationale for using probiotics in infectious diarrhoea is that they act against enteric pathogens by competing for available nutrients and binding sites, making the gut contents acid, producing a variety of chemicals, and increasing specific and non-specific immune responses. Probiotics reduced infectious diarrhoea in children and adults in various settings but a mechanism common to most probiotics, for example, colonization resistance, is effective against a wide range of gut pathogens.

Probiotic bacteria, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases. Probiotics have been studied extensively for their effects in preventing and treating a multitude of conditions, including the treatment of lactose intolerance, traveller's diarrhoea and the prevention and treatment of nosocomial diarrhoea. In acute diarrhoea, a reduction in the frequency of diarrhoeal symptoms has been reported in adults and children treated with probiotics. Among the beneficial microbes, Bifidobacterium is one of the best-known probiotic genus in the world, and it is widely applied in the dairy industry as a probiotic. Evidences from in vitro, in vivo, and clinical studies and long consumption history support the safety and health benefits of Bifidobacterium strains. The ingestion of yogurt fortified with B. longum reduced harmful bacteria such as Enterobacteriaceae, Streptococcus and C. perfringens, while at the same time alter the microbiota gut profile of volunteers with a significant increase of beneficial microbes Bifidobacterium and Lactobacillus species. Additionally, putrefactive substances in the intestinal environment were also reduced in the presence of the probiotic supplement. Such findings suggest that Bifidobacterium strains are safe and could be used further to evaluate its effect in preventing diarrhea and/or respiratory-related illness prevalence in young children.

Probiotic (Bifidobacterium infantis YLGB-1496) adheres to probiotic properties such as excellent tolerance to gastric acid, intestinal fluid and bile salt of the digestive system. Both probiotic and placebo products are manufactured under HACCP conditions. All products do not contain any animal-origin ingredients. The probiotic product contains probiotic and carrier while placebo contains only carrier. Sachets of products containing probiotic and placebo appear as light yellow powder. Both probiotic and placebo products are kept at storage temperature range below 30oC according to the condition recommended by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children (>12 months old, <7 years old).
* Having respiratory symptoms (having at least two of the following signs and symptoms: fever (even if only reported not measured), nasal obstruction, chills, sore throat, headache, cough, runny nose, olfactory disturbances, or taste disturbances; Pucarelli-Lebreiro et al., 2022).
* Healthy with current weight of P20-P80 percentile chart of children
* Infant formula powder does not contain probiotics; prebiotics FOS is not allowed, GOS <2g/ 100g is allowed
* Willing to commit throughout the experiment

Exclusion Criteria:

* Long term medication >6 months for any diseases
* Deformity
* Mothers with metabolic and/or chronic diseases
* Current or previous diseases, conditions or interventions that may interfere with the study (such as tolerance and/or growth and development), such as gastrointestinal malformations, chronic diarrhea, malabsorption syndromes, malnutrition, congenital immunodeficiency or surgery
* Oral antibiotics within 2 weeks before the intervention
* Nutritional supplements containing probiotics and prebiotics (except infant formula) within 2 weeks before the intervention
* Foods for special medical purposes or non-standard formula powders for lactose intolerance and galactosemia
* Probiotic allergies or possible food allergies (milk, etc.)
* Participated in other clinical studies 4 weeks before the intervention
* Unwilling to participate for any particular reason

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in children with respiratory tract infections upon administration of probiotic as assessed via pyrosequencing | 12-weeks
  Differences in microbiota abundance in fecal sample of children with respiratory tract infections upon administration o probiotic compared to placebo

SECONDARY OUTCOMES:
Clinical respiratory symptoms duration and frequency in children with respiratory tract infections upon administration of probiotic as assessed using the Monthly Health Questionnaire (as used in ClinicalTrials.gov (identifier number NCT02434042) | 12-weeks
  Changes in duration and frequency of respiratory illnesses symptoms from children on probiotic or placebo after 12-weeks, via the use of questionnaire.
Clinical gastrointestinal symptoms in children with respiratory tract infections upon administration of probiotic as assessed using the Monthly Gastrointestinal Questionnaire as used in ClinicalTrials.gov (identifier number NCT02434042) | 12-weeks
  Differences in duration and frequency of gastrointestinal symptoms of children upon administration of probiotic compared to placebo
Immunity profiles in children with respiratory tract infections upon administration of probiotic via the use of oral swabs | 12-weeks
  Differences in concentrations of proteins such as interleukins (IL-10, IL-4, IL-6, Tumour Necrosis Factor-alpha, Interferon gamma) in swab samples (ug/mL) of children upon administration of probiotic compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Adli Ali, MD, Principal Investigator — National University of Malaysia
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uma Mageswary M, Li P, Richmond RV, Azianey Y, Abd Hamid IJ, Taib F, Liong MT, Ali A, Tan JS, Zhang Y. Clinical benefits of Bifidobacterium infantis YLGB-1496 in modulating gut microbiota and immunity in young children. Front Nutr. 2026 Jan 5;12:1713135. doi: 10.3389/fnut.2025.1713135. eCollection 2025. PMID 41561177
- [Derived] Li P, Mageswary U, Ali A, Taib F, Koo TH, Yusof A, Jiang H, Lan H, Hung W, Liong MT, Zhang Y. Clinical effects of Bifidobacterium Longum Subsp. Infantis YLGB-1496 on children with respiratory symptoms. Front Nutr. 2025 Feb 19;12:1537610. doi: 10.3389/fnut.2025.1537610. eCollection 2025. PMID 40046755